CLINICAL TRIAL: NCT01598948
Title: Effect of Mipomersen on LDL-Cholesterol Levels in Patients With Severe LDL-Hypercholesterolemia and Atherosclerosis Treated by Regular LDL-Apheresis
Brief Title: Effect of Mipomersen on LDL-Cholesterol Levels in Patients Treated by Regular Apheresis
Acronym: MICA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ludwig-Maximilians - University of Munich (Other)
Responsible Party: Principal Investigator, Klaus Parhofer, Professor of Medicine, Ludwig-Maximilians - University of Munich
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MICA
Record Dates: First submitted 2012-05-12; First posted 2012-05-15 (Estimated); Last update posted 2015-09-02 (Estimated); Status verified 2015-09

CONDITIONS: Atherosclerosis; LDL-hypercholesterolemia
Keywords: hypercholesterolemia; apheresis; coronary heart disease; cerebrovascular disease; peripheral arterial disease
MeSH Terms: conditions — Atherosclerosis; Hypercholesterolemia; Coronary Disease; Cerebrovascular Disorders; Peripheral Arterial Disease | interventions — mipomersen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mipomersen (Experimental): Patients randomized to this arm will receive mipomersen 200 mg weekly
  Interventions: Drug: mipomersen
- Control (No Intervention): patients randomized to this arm will receive no additional drug

INTERVENTIONS:
Drug: mipomersen — mipomersen 200 mg subcutaneously every week for 37 weeks (phase 1: 26 weeks; phase 2: 11 weeks)
  Arms: Mipomersen

SUMMARY:
Elevated LDL-cholesterol is a major risk factor for heart disease. In patients with heart disease LDL-cholesterol should be lowered to levels below 70 mg/dl to prevent progression of disease. In most patients life style modification together with lipid lowering drug therapy is sufficient to achieve this goal. In some patients with severe forms of hypercholesterolemia, this may not be sufficient to reach goals and regular lipid apheresis (a costly and time intensive form of therapy) may be performed. Mipomersen is a new drug (apoB antisense oligonucleotide) that can lower LDL-cholesterol even in the most severe forms of LDL-hypercholesterolemia by 25-47%. It is unknown whether and to what extent mipomersen can decrease LDL-cholesterol in patients treated with regular apheresis. Phase 1 of the study will test how 6 months of weekly therapy with mipomersen affects LDL-cholesterol in patients with severe LDL-hypercholesterolemia treated with regular apheresis. Phase 2 will test in how many patients this will result in a meaningful reduction of apheresis time, apheresis frequency or if apheresis can be stopped completely.

ELIGIBILITY:
Inclusion Criteria:

* The patient fulfils German criteria for regular LDL-apheresis
* Regular (weekly) LDL-apheresis >/= 3 months
* The patient has fasting pre-apheresis LDL-C >/= 130 mg/dL at screening.
* The patient is receiving a stable, maximally tolerated, lipid-lowering regimen
* The patient has a body mass index (BMI) </= 40 kg/m2 with weight stable (± 4 kg) for > 6 weeks prior to screening.
* Written informed consent of the patient

Exclusion Criteria:

* The patient has experienced MI, percutaneous transluminal coronary intervention (PTCI), CABG, cerebrovascular accident, unstable angina, or acute coronary syndrome within 12 weeks of screening.
* The patient has insulin-dependent diabetes mellitus (Type 1), or if Type 2 diabetes, HbA1c > 8% at screening.
* The patient has New York Heart Association (NYHA) functional classification III or IV heart failure.
* The patient has systolic blood pressure > 160 mm Hg or diastolic blood pressure > 95 mm Hg at screening (despite antihypertensive medication/therapy).
* The patient has an active infection requiring systemic antiviral or antimicrobial therapy unless treatment expected to be completed by day 1.
* The patient has a positive test for HIV or hepatitis B or C at screening.
* The patient has any uncontrolled condition that may predispose to secondary hyperlipidemia such as uncontrolled hypothyroidism.
* The patient has had a malignancy within 5 years, except for basal or squamous cell carcinoma of the skin that has been adequately treated.
* The patient has clinically significant hepatic (e.g. History of confirmed non-alcoholic steatohepatitis NASH) or renal disease or Gilbert's syndrome.
* The patient has previously received mipomersen treatment.
* The patient is on chronic systemic corticosteroids or anabolic agents except for replacement therapy.
* The patient has received treatment with another investigational drug, biological agent, or device within 4 weeks of screening or 5 half-lives of the study agent, whichever is longer.
* The patient has a current or a recent history of drug or alcohol abuse, or unwillingness to limit alcohol consumption to within moderate limits (maximum 20 g alcohol per day and 80 g alcohol per week for males; maximum 10 g alcohol per day and 40 g alcohol per week for females).
* Patient not able to give consent.
* Patient without legal capacity who is unable to understand the nature, scope, significance and consequences of this clinical trial.
* Known history of hypersensitivity to the investigational drug or to drugs with a similar chemical structure
* Simultaneous participation in another clinical trial or participation in any clinical trial involving administration of an investigational medicinal product within 30 days prior to the beginning of the clinical trial.
* Patient with a physical or psychiatric condition which at the investigator's discretion may put the patient at risk, may confound the trial results, or may interfere with the patient's participation in this clinical trial
* Known or persistent abuse of medication, drugs or alcohol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-08; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in pre-apheresis LDL-cholesterol (phase 1 of the study) | 6 months
  pre-apheresis LDL-cholesterol concentration will be averaged from 3 subsequent aphereses (exactly 1 week apart) before initiation of mipomersen therapy and after 6 months of weekly apheresis therapy; apheresis conditions will not be changed.
Fraction of patients in whom apheresis conditions can be modified (phase 2 of the study) | 3 months
  In phase 2 of the study mipomersen will be given weekly. It will be evaluated in what fraction of patients this results in a decrease of apheresis time, apheresis frequency or stopping of apheresis.

SECONDARY OUTCOMES:
change in other lipid parameters | 6 months
  a number of additional lipid parameters will be evaluated before and during mipomersen therapy
Number of participants with adverse events | 9 months (phase 1 and 2 of the study)
Plasma concentrations of mipomersen | 4 days after injection
  pharmacokinetic sampling will be obtained following mipomersen administration at different time points during the study.

CONTACTS AND LOCATIONS:
Locations (1):
- University Munich, Munich, Germany